CLINICAL TRIAL: NCT02147470
Title: Evaluation of Renal Blood Flow Using Contrast Enhanced Ultrasound for Differential Diagnosis of Acute Kidney Injury in Cirrhotic Patients: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kambiz Kalantarinia, Associate Professor of Medicine, University of Virginia
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16603
Record Dates: First submitted 2013-12-17; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Liver Cirrhosis and Acute Kidney Injury
Keywords: cirrhosis of the liver; Acute kidney injury
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prerenal AKi, acute tubular necrosis and hepatorenal syndrome (Other): All subjects will undergo CEUS with the use of Definity to measure renal blood flow. At the same time clinical tools (urine output, response to volume expansion, urine sodium, urine output, fractional excretion of sodium and urea and urine microscopy) will be used to differentiate between prerenal AKI, ATN and HRS. the quantity and patterns of RBF measured by CEUS will be compared between these three groups.
  Interventions: Drug: Definity ultrasound contrast agent

INTERVENTIONS:
Drug: Definity ultrasound contrast agent — All subjects will undergo CEUS of the kidney at baseline to measure renal blood flow. This procedure will be repeated after volume expansion and if indicated, once again after treatment with albumin, midodrine and octreotide.
  Other Names: Contrast Enhanced Ultrasound using Definity

SUMMARY:
Hepatorenal syndrome (HRS) is a common cause of acute kidney injury (AKI) in cirrhotic patients and has a one month survival rate of 50% and a 3 month survival rate of 20%. The leading theory behind HRS is selective vasoconstriction of renal vasculature in the setting of decreased systemic vascular resistance. Patients with liver cirrhosis suffer from a large degree of third spacing in the form of peripheral edema and ascites. In addition treatment with multiple drugs, including diuretics puts these patients at higher risks of prerenal AKI and ischemic acute tubular necrosis (ATN). AKI occurring due to HRS, prerenal AKI and ischemic or nephrotoxic ATN have different pathophysiologic mechanisms and are treated differently with significantly different outcomes. While renal perfusion is expected to be reduced in HRS and prerenal AKI, it is normal or increased in ATN. Prerenal AKI has the most favorable prognosis among these pathologies and treatment simply consists of volume expansion with blood, albumin, crystalloids or colloids. In clinical practice vasoactive agents such as midodrine and octreotide are used to increase the tone of splanchnic vessels and to improve renal perfusion. These interventions would not affect renal function in cases with ATN. Unfortunately, the diagnostic criteria proposed by the International Club for Ascites (ICA) for HRS are not specific and do not always exclude patients with other forms of acute kidney injury. Therefore, availability of a simple diagnostic tool for measurement of renal blood flow (RBF) at the bedside would be of great value in management of cases with cirrhosis of the liver presenting with acute reduction in kidney function. However, currently, there are no practical and simple tools available for this purpose.

Contrast enhanced ultrasonography (CEU) involves the intravenous injection of gas-filled microbubbles to enhance the ultrasound image of the organs and mainly to assess tissue vascularity and blood flow. We and others have used CEU to assess changes in RBF in response to physiologic stimuli and therapeutic interventions. Here we propose a prospective, pilot diagnostic study to validate the use of CEU, in assessing RBF in cirrhotic patients with AKI, and to assess the utility of CEU to differentiate between causes of AKI in cirrhotic patients.

Our hypothesis is that CEU will show arteriolar vasoconstriction and decreased blood flow in the renal cortex in patients with HRS which would not change in response to volume expansion. On the contrary, patients with prerenal AKI will have reduced RBF which will increase after volume expansion. Finally, those with ATN will not have a reduced RBF at baseline.

We plan to enroll 25 patients with liver cirrhosis and acute kidney injury who are admitted to the University of Virginia hospital into the study.

CEU will be performed on all subjects to measure baseline RBF. CEU will be repeated in all subjects within 24 hours after volume expansion with at least 1gm/kg of albumin (up to 100 gm/day) to assess a potential change. Hourly urine output and serum creatinine will be monitored for potential renal response to the volume expansion as part of clinical care. For the subgroup of subjects who receive treatment with combination therapy with albumin, midodrine, and octreotide (AMO) RBF assessment with CEU will be repeated after at least 48 hours of receiving this combination. Renal response will be assessed by monitoring urine output and serum creatinine monitored as part of clinical care. All subjects will have measurements of fractional excretion of sodium (FENa) and urea (FEUrea) and urine microscopy as a part of their routine clinical care (work up of AKI). The results of these tests and the response to volume expansion will be used to categorize subjects into three categories of AKI (HRS, prerenal AKI, ATN). Correlations between RBF and its changes between different therapeutic interventions and renal diagnosis will be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Cirrhosis of liver
* Hospitalization at University of Virginia Medical Center
* Diagnosis of acute kidney injury based on AKIN criteria

Exclusion Criteria:

* Known history of a right to left intracardiac shunt
* Known history of pulmonary hypertension, including portopulmonary hypertension
* Pregnancy or lactation
* History of allergies to Definity®
* History of Liver or Kidney Transplant
* Patient on hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To assess the utility of monitoring of RBF using CEU in management of AKI in patients with liver cirrhosis. | 24 - 48 hours

SECONDARY OUTCOMES:
Pattern of blood flow distribution in the kidney in different cases of AKI | 0 - 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States